CLINICAL TRIAL: NCT04448704
Title: Understanding the Mental Health of Migrant Workers During the COVID-19 Outbreak
Status: Completed | Type: Observational
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Other Study IDs: CCF@EXPO/R001/2020
Record Dates: First submitted 2020-06-25; First posted 2020-06-26 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Mental Health Issue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the mental health impact of the COVID-19 pandemic on international migrant workers by (1) documenting mental health symptoms among migrant workers and (2) identifying risk and protective factors during the pandemic.

DETAILED DESCRIPTION:
Worldwide, there are an estimated 164 million migrant workers. Although studies have documented how migrant workers have an increased risk of adverse mental health outcomes, little is known about their mental health burden during a large-scale health crisis.

In the current COVID-19 outbreak, migrant workers represent 9 in 10 of the COVID-19 cases in Singapore, with 25 dormitories gazetted to contain the spread of the virus. Correspondingly, these measures have placed a spotlight on the mental well-being of migrant workers.

In this research protocol, the investigators propose to administer a survey to understand the prevalence and predictors of mental health symptoms amongst migrant workers in Singapore. In particular, prior meta-analyses have identified COVID-19 health concerns, quarantine status, financial instability, exposure to news and misinformation and demographics (i.e., gender, age, education) as risk factors for poor mental health amongst the general population. By assessing these factors amongst the migrant worker population and documenting their impact on migrant workers' mental health, we hope to identify workers in greatest need of support during the ongoing pandemic and provide empirical evidence to guide public health policies.

ELIGIBILITY:
Inclusion Criteria:

* ≥21 years of age
* Hold a government-issued work permit identifying employment status

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Migrant workers employed in manual labor jobs within Singapore
Sampling Method: Non-Probability Sample
Enrollment: 1011 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2020-10-11 (Actual); Study Completion 2020-10-11 (Actual)

PRIMARY OUTCOMES:
DASS-21 Scores | single measurement upon study enrolment
  Depression, Anxiety and Stress Scale (DASS-21) is a validated 21-item measure that has been widely used during the current COVID-19 pandemic.

CONTACTS AND LOCATIONS:
Locations (1):
- EXPO, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No